CLINICAL TRIAL: NCT06090136
Title: A Study Evaluating Safety and Pharmacokinetics of a Single Oral TPN171H in Elderly Subjects
Brief Title: Safety and Pharmacokinetics of a Single Oral TPN171H in Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPN171H-06
Record Dates: First submitted 2023-06-21; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TPN171H (Experimental): 5 mg TPN171H tablets，single dose,oral
  Interventions: Drug: TPN171H

INTERVENTIONS:
Drug: TPN171H — 5 mg TPN171H tablets，single dose,oral

SUMMARY:
It is a single-center, open-label, Phase I clinical study evaluating the safety and pharmacokinetics of a single oral TPN171H in elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 65 years old；
2. Male≥50kg，femal≥45kg, Body mass index should be between 18 and 30 kg/m2 (inclusive)；
3. No major organ dysfunction；normal heart, liver and kidney function;
4. Physical examination, vital signs examination, laboratory examination (blood routine, urine routine, blood biochemistry), 12 lead ECG, Abdominal ultrasound, chest X-ray results were normal or abnormal but investigator judged suitable for participating in this trial;
5. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the written informed consent

Exclusion Criteria:

1. Allergies to test preparations, any of their ingredients, and related preparations; With allergies or allergic diseases;
2. Surgical condition or condition that may significantly affect ADME of the drug, urgical condition or condition that may pose a hazard if the subject participating in the study
3. Myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass grafting, congestive heart failure, severe arrhythmias, cerebrovascular accidents, including transient ischemic attack within 3 months before inclusion;
4. Taken any of drugs(Inhibits or induces liver metabolism) within 2 weeks before inclusion；administered with Nitrate/Nitric oxide (NO) donors。
5. With a history of the following ocular diseases: nonvascular anterior ischemic optic neuropathy (NAION), abnormal color vision, hereditary retinopathy (e.g. Retinitis pigmentosa), and macular degeneration；
6. A history of sudden decrease or loss of hearing；
7. A history of postural hypotension；
8. Blood loss ≥400 mL within 3 months before inclusion；
9. Participated in other drug clinical trials or medical devices clinical trials within 3 months before administration；
10. Drink alcohol at least 2 times a day or more than 14 times a week in the 6 months prior to enrollment or alcoholics(Drink alcoholics defined as 125 mL of wine, 220 mL of beer, or liquor50mL； Alcoholism is defined as 5 or more drinks in approximately 2 hours) ;
11. A history of drug use or have been screened positive for drug abuse;
12. Smoked more than 10 cigarettes a day within 6 months prior to inclusion;
13. hepatitis B surface antigen (HBsAg),hepatitis C virus antibody,treponema pallidum antibody,Human immunodeficiency virus antibody (HIV)positive;
14. Other factors that the investigator considered inappropriate for the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Adverse events | 7 days after dosing
  Number of Participants With treatment-related Adverse Events and Serious Adverse Events
Pharmacokinetic parameter of TPN171H:Tmax | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:Tmax
Pharmacokinetic parameter of TPN171H:Cmax | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:Cmax
Pharmacokinetic parameter of TPN171H:T1/2 | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:T1/2
Pharmacokinetic parameter of TPN171H:AUC0-t | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:AUC0-t
Pharmacokinetic parameter of TPN171H:AUC0-∞ | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:AUC0-∞
Pharmacokinetic parameter of TPN171H:AUC0-24h | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:AUC0-24h
Pharmacokinetic parameter of TPN171H:Ke | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:Ke
Pharmacokinetic parameter of TPN171H:Vd | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:Vd
Pharmacokinetic parameter of TPN171H:MRT | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:MRT
Pharmacokinetic parameter of TPN171H:CL/F | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:CL/F
Pharmacokinetic parameter of TPN171H:BRPP | 48 hours after dosing
  Pharmacokinetic parameter of TPN171H:BRPP

CONTACTS AND LOCATIONS:
Overall Officials: Gangyi Liu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No